CLINICAL TRIAL: NCT06054256
Title: Efficacy of Digitally Delivered and Face-to-face Group Cognitive Behavioural Therapy for Insomnia in Pregnant Women With Comorbid Insomnia and Depression: A Randomised Controlled Trial
Brief Title: Effects of Digitally Delivered and Group-based CBT-I in Pregnant Women With Comorbid Insomnia and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Stanford University (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA220035
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related; Depression; Insomnia
Keywords: Depression; Insomnia; Antenatal; Cognitive behavioural therapy; Pregnancy
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group CBT-I (Experimental): The group CBT-I will receive 6-session group-based CBT-I.
  Interventions: Behavioral: Group CBT-I
- App-based CBT-I (Experimental): The app-based CBT-I group will receive 6-session CBT-I via smartphone.
  Interventions: Behavioral: App-based CBT-I
- Health-related psychoeducation control (Sham Comparator): The control group will receive group-based health-related psychoeducation, a format that has been adopted in the previous research, in order to provide the credibility of the intervention to the participants, and to control for the potential effects of attention and nonspecific components, e.g., receiving health-related information, expectations of benefit. It will also consist of 6 weekly sessions which contain education on healthy diet, exercise habits, sleep hygiene and self-care specific to pregnancy, but will not include any active therapeutic components of CBT-I.
  Interventions: Other: Health related psychoeducation

INTERVENTIONS:
Behavioral: Group CBT-I — The group-based intervention will consist of 6 weekly sessions (90-min, 5-8 pregnant women in each group). The treatment components aim to address the behavioural, cognitive and physiological factors perpetuating insomnia with the followings: psycho-education about sleep and sleep hygiene (e.g., psychoeducation about sleep during pregnancy and normal development and patterns of infant sleep, psychoeducation on ways of improving infant sleep, strategies to limit the development of unwanted sleep associations, etc.), stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Arms: Group CBT-I
Behavioral: App-based CBT-I — The smartphone app-based intervention will consist of 6 weekly sessions. The app-based intervention will involve a self-paced, fully automated digital programme with interactive components. The structure of the app involves six sequential modules (comparable to the six treatment sessions delivered in groups) with different elements to engage the users, such as animated videos, case vignettes, narration, quizzes, and homework assignment. Each module will be unlocked and released to the participants every week after the previous module has been completed. Personalised feedback will be provided by the app following the completion of sleep diary each week. Automated messages will be sent to the participants regularly via phone to remind them of implementing learned strategies after each module, as well as timely completing the treatment modules and sleep diaries.
  Arms: App-based CBT-I
Other: Health related psychoeducation — The control group will receive 6 sessions of group-based health-related psychoeducation, a format that has been adopted in the previous research, in order to provide the credibility of the intervention to the participants, and to control for the potential effects of attention and nonspecific components.
  Arms: Health-related psychoeducation control

SUMMARY:
Major depressive disorder (MDD) is a debilitating and recurrent illness associated with a constellation of grave consequences and is among the most common psychiatric disorders during the pregnancy and postpartum periods. Meanwhile, sleep disturbance, particularly insomnia, is among the most prevalent and prominent presenting complaints in pregnant women with depression. Despite its high prevalence, insomnia often remains overlooked and under-treated in clinical practice. However, growing evidence suggests an intricate relationship between insomnia and depression, which has become an area in need of further focused attention. The optimal treatment for managing both antenatal depression and insomnia remains controversial. Only few pilot studies have evaluated the effects of cognitive behavioural therapy for insomnia (CBT-I) for antenatal insomnia. Whilst face-to-face CBT-I has shown the promise in managing insomnia in pregnant women, several barriers to implementation remain in clinical practice (e.g., a lack of trained therapists, long waiting time). Pregnant women also face additional unique barriers to obtaining insomnia treatment, including having other recurring prenatal health appointments, limitations in mobility or transportation, and financial concerns. There is growing evidence supporting the feasibility and comparable efficacy of digital CBT-I (effect size Cohen's d ranging from 0.69 to 0.8) as compared to a control intervention (e.g., sleep hygiene education, relaxation) for treating adult insomnia. However, little is known about the effects of different treatment modalities (group-based vs. app-based CBT-I) during pregnancy. This study aims to conduct a randomised controlled trial to examine the effects of group-based CBT-I and smartphone app-based CBT-I as compared to health education control condition in pregnant women with comorbid depression and insomnia on improving maternal sleep and depressive symptoms, other clinical and daytime symptoms, and overall functional improvement, as well as mother-infant-relationship.

DETAILED DESCRIPTION:
A randomised parallel-group controlled trial will be conducted in pregnant women with comorbid insomnia and depression. Eligible subjects will be randomised to one of the following groups: group-based CBT-I + Usual care (UC), app-based CBT-I + UC, or health education + UC. Randomization will be performed using stratified blocked randomization, stratified by the severity of insomnia at baseline. Assessments will be conducted at baseline and post-treatment (week 6/at the conclusion of last session). Subjects will be also assessed for their sleep and mood symptoms at week 2/at the conclusion of session 2 and week 4/at the conclusion of session 4. Subjects in the control group will be offered CBT-I after post-intervention follow-up. Additional assessments will be conducted in the two active treatment groups at postpartum 3-month and 6-month. A further follow-up assessment will be scheduled at 12-month postpartum to particularly examine whether intervention effects can sustain over time in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above;
2. 28-32 weeks of gestation at the entry of the study;
3. Having a DSM-5 diagnosis of insomnia disorder and with a score on Insomnia Severity Index (ISI) ≥8;
4. Having a DSM-5 diagnosis of depressive disorder as confirmed by the M.I.N.I. International Neuropsychiatric Interview (MINI) and with mild to moderate depressive symptoms (an Edinburgh Postnatal Depression Scale (EPDS) score ≥7 and ≤19);
5. Singleton pregnancy;
6. Being capable of providing informed consent.

Exclusion Criteria:

1. Having a health-related high-risk factor, e.g., high blood pressure, diabetes, being HIV-positive, uncontrolled thyroid or seizure disorder;
2. Having a clinically diagnosed sleep disorder (e.g., obstructive sleep apnoea, periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep-wake disorders, parasomnias) based on the Diagnostic Interview for Sleep Patterns and Sleep Disorders (DISP), a validated semi-structured clinical interview for assessing major sleep disorders according to ICSD-2 criteria;
3. Having a significant mental health condition, including posttraumatic stress disorder (current), panic disorder if associated with nocturnal panic attacks > 4 times in the past month, bipolar disorders, psychotic disorders, substance use disorders (during pregnancy);
4. The subject, in the opinion of the investigator, has a significant risk of suicide, or has a suicidality level rated as moderate or above in the MINI Suicidality Module;
5. Concurrent, regular use of medications or substance known to directly affect sleep quality and continuity (e.g., hypnotics, melatonin, steroids);
6. Initiation of or change in antidepressant medication within past 2 months;
7. Ongoing pharmacologic or nonpharmacologic treatments for insomnia;
8. Night shift worker;
9. With hearing or speech deficit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of insomnia symptoms | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at the conclusion of session 2 and 4, postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Insomnia Severity Index (ISI) is a self-rated scale to assess the severity of insomnia symptoms. Possible scores range from 0 to 20, with higher scores indicating greater insomnia severity.
Change of depressive symptoms | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at the conclusion of session 2 and 4, postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report questionnaire used to assess the severity of depressive symptoms during both prenatal and postnatal periods. Possible scores range from 0 to 30, with higher scores indicating more serious depressive symptoms.

SECONDARY OUTCOMES:
Change of pregnancy anxiety | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2) is a 10-item self-report inventory to assess pregnancy anxiety. Possible scores range from 10 to 50, with higher scores indicating more serious pregnancy anxiety.
Change of pregnancy stress | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Pregnancy Stress Rating Scale (PSRS) is a 36-item scale to measure psychological stress felt by women using a 5-point scale, ranging from never (1 point) to very extreme (5 points). A higher score indicates a higher stress level.
Change of self-report emotional states of depression, anxiety and stress | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Depression Anxiety Stress Scales (DASS-21) consists of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS scales contains 14 items. Higher scores suggest more depression, anxiety and stress, respectively.
Change of suicidal ideation | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of sleep quality | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of sleep diary measure (time in bed, TIB) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours.
Change of sleep diary measure (total sleep time, TST) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours.
Change of sleep diary measure (sleep onset latency, SOL) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins.
Change of sleep diary measure (wake after sleep onset, WASO) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins.
Change of sleep diary measure (sleep efficiency, SE) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %.
Change of objective sleep measure (time in bed, TIB) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours.
Change of objective sleep measure (total sleep time, TST) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours.
Change of objective sleep measure (sleep onset latency, SOL) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins.
Change of objective sleep measure (wake after sleep onset, WASO) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins.
Change of objective sleep measure (sleep efficiency, SE) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %.
Change of dysfunctional beliefs and attitudes about sleep | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change of pre-sleep arousal | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Pre-Sleep Arousal Scale (PSAS) is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.
Change of sleep reactivity | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Ford Insomnia Response to Stress Test (FIRST) consists of 9 items designed to measure sleep reactivity. Possible scores range from 9 to 36. A higher score indicates higher sleep activity.
Change of sleep hygiene and practice | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Sleep Hygiene Practice Scale (SHPS) is a 30-item self-rated scale measuring sleep hygiene behaviors, ranging in total scores from 30 to 180, with higher scores indicating lower levels of sleep hygiene.
Change of daytime sleepiness | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Epworth Sleepiness Questionnaire (ESS) is used to measure self-reported excessive daytime sleepiness (EDS). The total score of ESS ranges from 0 to 24, with higher scores indicating higher daytime sleepiness.
Change of subjective cognitive performance | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Cognitive Failures Questionnaire (CFQ) is a 20-item self-rated scale measuring perceived failures in daily cognitive tasks. Possible total scores range from 0 to 80, with higher scores indicating higher cognitive failures.
Change of daytime fatigue | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change of quality of life | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  The Short Form 12 (SF-12) Health Related Quality of Life (HRQL) is a 12 item self-reported questionnaire to measure health related quality of life. A higher score on SF-12 represents a better health-related quality of life.
Change of postpartum mother-infant-relationship | Postpartum 3-month, 6-month and 12-month for those in the two active treatment groups.
  Mother-Infant Bonding Questionnaire (MIBQ) is a 8 item self-reported scale to assess maternal bonding of mothers with their babies during the postpartum period. Total scores range from 0 to 24. A high score indicates worse mother-to-infant bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No